CLINICAL TRIAL: NCT01828567
Title: Will Veterans Engage in Prevention After HRA-guided Shared Decision Making?
Acronym: ACTIVATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CRE 12-288
Record Dates: First submitted 2013-04-05; First posted 2013-04-10 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Health Risk Appraisal; Heart Disease; Prevention
Keywords: veterans; health risk assessment; primary prevention; shared decision making; Healthy Living Assessment
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Primary care phone-based prevention coaching using shared decision making following a Healthy Living Assessment
  Interventions: Behavioral: Shared decision making with a Prevention Coach
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Shared decision making with a Prevention Coach — A series of two phone sessions with a prevention coach. The first to engage the veteran to choose a preferred prevention program and link them to Patient Aligned Care Team (PACT), and a follow-up call one month later to assess the progress of the prevention plan.
  Arms: Intervention

SUMMARY:
The VA has committed to disseminate a web-based Healthy Living Assessment(HLA) tool and use it as the cornerstone of a personalized prevention plan to engage patients to improve their health behaviors that lead to high health risk. Health risk assessments done in isolation, however, do not generally lead to behavior change. Our study will test the effectiveness of a Shared Decision Making intervention designed to activate Veterans to enroll in effective prevention programs. The intervention will be conducted over the telephone, by a prevention coach, and will be linked to the patients' primary care team. The co-primary outcomes will be patient activation and patient enrollment in prevention programs; 10-year risk of major cardiac events will also be measured.

DETAILED DESCRIPTION:
Over half of all deaths, and many illnesses, can be attributed to four modifiable risk factors: tobacco use, overweight/obesity, physical inactivity, and alcohol use. There are clear links between these modifiable factors and heart disease, cancer, chronic lung disease, and stroke which continue to be the leading causes of death in the United States. Significant improvements have been made in controlling conditions that lead to heart disease, cancer and stroke (e.g., hypertension and hyperlipidemia). However, the underlying behavioral factors (e.g., obesity, tobacco use, and physical inactivity) have not been addressed as well. Prevention is particularly important for Veterans because of the high prevalence of significant risk factors for poor health. For example, more than 70% of Veterans Health Administration (VHA) patients are overweight (body mass index [BMI] 25kg/m2) and one-third are obese (BMI 30kg/m2), which is significantly higher than the US population. Smoking also remains a significant problem among Veterans, with VHA enrollment data from 2010 indicating a prevalence of 20%. Younger Veterans are at particularly high risk for developing chronic illnesses because they are more likely to be overweight/obese and smoke more heavily than non-Veterans.

The investigators propose a two-site, two-arm randomized trial measuring the effectiveness of a Shared Decision Making (SDM) intervention in activating Veterans to enroll in effective prevention services, and improve cardiovascular risk, compared to Veterans Administration (VA) usual care. The study will be performed at the Durham and Ann Arbor Veterans Administration Medical Centers (VAMCs). Each arm will have 225 patients; patients will be VA users with at least one modifiable risk factor (obese, inactive, or tobacco user) who are not currently enrolled in a prevention service. The SDM intervention will be conducted by a prevention coach, telephone based, and will use the output from VHA's Healthy Living Assessment (HLA) to engage Veterans in a conversation where individual preferences are matched to behaviors, and choices for specific prevention services. The resulting prevention action plan will be shared with the Veterans primary care team, and documented in the medical record.

Outcomes will be obtained at baseline, 1 month and 6 months after enrollment by blinded research personnel. The primary outcomes will be: 1) proportion enrolled in effective prevention services; and 2) change in the Patient Activation Measure (PAM). The secondary outcome is 10-year risk of coronary events, as measured by Framingham Risk Score (FRS). Process evaluations of the intervention and its implementation will also be conducted to inform future dissemination and implementation should it prove effective.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, patients must meet the following:

* enrolled in primary care at the Durham or Ann Arbor Health Care Systems
* have one modifiable risk factor identified by a healthy living assessment (physical inactivity, overweight or obese by BMI, or tobacco user)

Exclusion Criteria:

Individuals will be excluded if they have any of the following:

* have been hospitalized for a stroke, myocardial infarction or coronary artery revascularization in the past three months
* have an active diagnosis of psychosis
* have any other health condition they feel would impede participation in the study
* reside in a nursing home
* are severely impaired in hearing or speech, so that they cannot respond to telephone calls
* have significant cognitive or memory impairment
* do not have access to a telephone
* are participating in another prevention intervention study
* are already enrolled in a formal prevention service

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Z. Oddone, MD MHSc, Principal Investigator — Durham VA Medical Center, Durham, NC; Laura J. Damschroder, MPH, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared. Final data sets will be maintained locally until enterprise-level resources become available for long-term storage and access. Guidance on request and distribution processes will be provided by ORD.
  A local privacy officer and study statistician will certify that the dataset contains no PHI prior to distribution. Data will be provided to requestor in electronic form.

REFERENCES:
- [Result] Oddone EZ, Damschroder LJ, Gierisch J, Olsen M, Fagerlin A, Sanders L, Sparks J, Turner M, May C, McCant F, Curry D, White-Clark C, Juntilla K. A Coaching by Telephone Intervention for Veterans and Care Team Engagement (ACTIVATE): A study protocol for a Hybrid Type I effectiveness-implementation randomized controlled trial. Contemp Clin Trials. 2017 Apr;55:1-9. doi: 10.1016/j.cct.2017.01.007. Epub 2017 Jan 24. PMID 28126455
- [Result] Oddone EZ, Gierisch JM, Sanders LL, Fagerlin A, Sparks J, McCant F, May C, Olsen MK, Damschroder LJ. A Coaching by Telephone Intervention on Engaging Patients to Address Modifiable Cardiovascular Risk Factors: a Randomized Controlled Trial. J Gen Intern Med. 2018 Sep;33(9):1487-1494. doi: 10.1007/s11606-018-4398-6. Epub 2018 May 7. PMID 29736750
- [Derived] Olsen MK, Stechuchak KM, Hung A, Oddone EZ, Damschroder LJ, Edelman D, Maciejewski ML. A data-driven examination of which patients follow trial protocol. Contemp Clin Trials Commun. 2020 Aug 13;19:100631. doi: 10.1016/j.conctc.2020.100631. eCollection 2020 Sep. PMID 32913914
- [Derived] Sloan C, Stechuchak KM, Olsen MK, Oddone EZ, Damschroder LJ, Maciejewski ML. Short-Term VA Health Care Expenditures Following a Health Risk Assessment and Coaching Trial. J Gen Intern Med. 2020 May;35(5):1452-1457. doi: 10.1007/s11606-019-05455-z. Epub 2020 Jan 2. PMID 31898118
- [Derived] Nouri SS, Damschroder LJ, Olsen MK, Gierisch JM, Fagerlin A, Sanders LL, McCant F, Oddone EZ. Health Coaching Has Differential Effects on Veterans with Limited Health Literacy and Numeracy: a Secondary Analysis of ACTIVATE. J Gen Intern Med. 2019 Apr;34(4):552-558. doi: 10.1007/s11606-019-04861-7. Epub 2019 Feb 12. PMID 30756302

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Primary care phone-based prevention coaching using shared decision making following a Healthy Living Assessment
  Shared decision making with a Prevention Coach: A series of two phone sessions with a prevention coach. The first to engage the veteran to choose a preferred prevention program and link them to PACT, and a follow-up call one month later to assess the progress of the prevention plan.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 208 | 209
1 Month | 172 | 192
Completed | 177 | 199
Not Completed | 31 | 10
Not completed — Lost to Follow-up | 27 | 9
Not completed — Excluded - did not meet criteria | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 208 | 209 | 417
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (12.7) | 56.3 (11.7) | 55.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 25 | 61
  Male | 172 | 184 | 356
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 90 | 79 | 169
  White | 99 | 110 | 209
  Other | 19 | 20 | 39
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 208 | 209 | 417

OUTCOME MEASURES:

1. Primary Outcome: Enrollment in Prevention Services
Description: Proportion of veterans enrolled in effective prevention services including weight loss, healthy eating, physical activity, and smoking cessation programs.
Time Frame: 1 and 6 months (cumulative)
Population: Unknowns were removed from the denominator: Intervention n=29; control n=15.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 179 | 194
participants | 91 | 56
Statistical Analysis 1: Comparison: Intervention vs Control; The first primary outcome is the cumulative enrollment in prevention programs over the six months of follow up. This will be assessed via self-report at months 1 and 6. As defined by the eligibility criteria, all patients will have a value of 0 at baseline; Test type: Other — A logistic regression model was used. The null hypothesis is that there is no difference in improvement prevention program enrollment between the usual care and intervention arms by month 6; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.54, 95% CI 2-sided [1.66 to 3.89]

2. Secondary Outcome: Patient Activation Measures (PAM)
Description: Patient Activation Measures (PAM) assesses patients capacity to manage their health. Improvement in PAM scores indicate responsiveness to interventions and improvements in self-management behaviors. Minimum score is a zero and maximum is one hundred. Higher score is better. The protocol specifies co-primary outcomes with enrollment in prevention services specified as the most clinically relevant
Time Frame: Baseline assessment
Measure: Mean (Standard Deviation); unit: average score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 208 | 209
average score | 62.4 (12.7) | 60.6 (12.3)

3. Secondary Outcome: Patient Activation Measures
Description: as for outcome 2
Time Frame: 1 month assessment
Measure: Mean (Standard Deviation); unit: average score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 172 | 192
average score | 63.7 (13.8) | 61.4 (11.1)
Statistical Analysis 1: Comparison: Intervention vs Control; For the primary hypothesis we will be examining the effect during the 1-month long intervention delivery period; Test type: Other; p = 0.204, Repeated Measures — A general linear model with an unstructured covariance matrix to take into account the within-patient correlation between repeated measures over time; This model assumes the groups have equal baseline means; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-0.8 to 3.7] — We estimate the parameters in the model using the SAS procedure MIXED (SAS Version 9.4, Cary, NC). The null hypothesis is that there is no difference in improvement in PAM scores between the usual care and intervention arms at 1 month

4. Secondary Outcome: Patient Activation Measures
Description: as for outcome 2
Time Frame: 6 months assessments
Measure: Mean (Standard Deviation); unit: average score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 177 | 199
average score | 67.0 (13.0) | 63.2 (13.3)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Equivalence — This model assumes the groups have equal baseline means, which is appropriate for a randomized controlled trial and is equivalent in efficiency to an ANCOVA model; p = 0.030, Repeated Measures — A general Linear model with an unstructured covariance matrix to take into account the within-patient correlation between repeated measures over time. For the primary hypothesis we will be assessing sustainability at 6 months; This model assumes the groups have equal baseline means; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [0.2 to 4.7] — We estimate the parameters in the model using the SAS procedure MIXED (SAS Version 9.4, Cary, NC). The null hypothesis is that there is no difference in improvement in PAM scores between the usual care and intervention arms at 6 month

5. Secondary Outcome: Framingham Risk Score
Description: The Framingham Risk Score is a gender-specific algorithm used to estimate the 10-year cardiovascular risk of an individual. This is not a scale however, lower score indicates less risk.
Time Frame: Baseline
Population: Unknowns were removed from the denominator: Intervention n=7; control n=2.
Measure: Mean (Standard Deviation); unit: average score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 201 | 207
average score | 21.8 (16.8) | 22.7 (16.8)

6. Secondary Outcome: Framingham Risk Score
Description: as for outcome 5
Time Frame: 6 months
Population: Unknowns were removed from the denominator: Intervention n=22; control n=18.
Measure: Mean (Standard Deviation); unit: average score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 155 | 181
average score | 22.4 (17.5) | 22.5 (16.3)
Statistical Analysis 1: Comparison: Intervention vs Control; Our secondary outcome of interest is the Framingham Risk Score, measured at baseline and month 6; Test type: Equivalence — This model assumes the groups have equal baseline means; p = 0.330, Repeated Measures; A general linear model with an unstructured covariance matrix to take into account the within-patient correlation between repeated measures over time; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-0.7 to 2.2] — We estimate the parameters in the model using the SAS procedure MIXED (SAS Version 9.4, Cary, NC). The null hypothesis is that there is no difference in improvement in FRS scores between the usual care and intervention arms at 6 month

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months.
Description: Adverse events information was collected from participants if they reported events at the 1 month and 6 month outcome assessments. Adverse event information was also collected from patients through contact with the coach interventionist or if during updating of clinical records it was discovered that an adverse event had occurred with a patient. Adverse events were monitored/assessed without regard to the specific Adverse Event Terms.
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 65/208 | 53/209
Other Adverse Events (participants affected / at risk) | 0/208 | 0/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=208) | Control (N=209)
Study Safety Protocol (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hospitalization (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Study Safety Protocol (Cardiac disorders) | 4 (4) | 2 (2)
Hospitalization (Cardiac disorders) | 2 (2) | 0 (0)
Important Medical Event (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization (Endocrine disorders) | 0 (0) | 1 (1)
Hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hospitalization (General disorders) | 1 (1) | 0 (0)
Hospitalization (Hepatobiliary disorders) | 2 (2) | 0 (0)
Protocol Deviation (Investigations) | 45 (45) | 36 (36)
Hospitalization (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Emergency Room Visit (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Important Medical Event (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Important Medical Event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Hospitalization (Psychiatric disorders) | 5 (5) | 2 (2)
Important Medical Event (Psychiatric disorders) | 1 (1) | 0 (0)
Emergency Room Visit (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Important Medical Event (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization (Surgical and medical procedures) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes